CLINICAL TRIAL: NCT03666403
Title: Department of Pediatrics, Taipei Veterans General Hospital, Taipei, Taiwan
Brief Title: Airway Pressure and Lumen Changes During NIV With Flexible Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-07-009B
Record Dates: First submitted 2018-08-28; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Airway Disease
Keywords: airway pressure; bronchomalacia; tracheomalacia; positive pressure ventilation; airway expansion; noninvasive ventilation
MeSH Terms: conditions — Bronchomalacia; Tracheomalacia

STUDY DESIGN:
Intervention Model Description: Upon the pharyngeal oxygen setting, this classic NIV operation was performed as per our protocol illustrated in the following steps. Firmly closed the mouth, then intermittently applied: a) assisted inspiration by nose-closure accompanied with cricoid depression; and b) assisted expiration by the release of above nose and cricoid maneuver, and simultaneous doing abdomen-compression. The above assisted ventilation cycle was performed at a rate of 0-20 cycles per minute. The bronchoscopist optionally executed both the FB and the nose- closure and release, whereas an assistant delivered the abdomen-compression.
Masking Description: Three modes with different ventilation (nose-close) rates were studied: mode A, spontaneous breathing, with only PhO2 support, no rate; mode B, rate of 15-20 per minute with Ti 1.0 seconds; and mode C, rate of 5-10 per minute with Ti 2-4 seconds. During FB, every patient underwent all these three modes sequentially, from A to C. When the oxygen desaturation (<90%) or bradycardia (<100 beat/min) persisted more than 10 seconds, the FB was terminated. After the child was stabilized, FB was resumed, starting from the nose-close, but shifted to the next mode of NIV support. When the mode C still failed to maintain an acceptable vital status, the FB procedure was aborted with the removal of the bronchoscope to allow more aggressive NIV or even traditional resuscitation technique including endotracheal intubation and manual ventilation with high FiO2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): This prospective one-year study enrolled consecutive 30 children of ≤3 years-old with suspected major airway diseases and therefore scheduled for diagnostic FB. During FB, PIP measurements and associated lumen images were obtained at six airway locations using three studied NIV modes, including 1) NIV rate: 0/min, 2) NIV rate: 10-20/min, 3) NIV rate: 5-10/min.
  Interventions: Procedure: NIV rate: 0/min; Procedure: NIV rate: 10-20/min; Procedure: NIV rate: 5-10/min

INTERVENTIONS:
Procedure: NIV rate: 0/min — A basic PhO2 flow was routinely provided. A small pharyngeal catheter with warmed, humidified and fixed pure oxygen flow was inserted via one nostril to ensured catheter tip positioning in the oropharynx. The NIV was performed in the following steps. Firmly closed the mouth, then intermittently applied a) assisted inspiration by nose-closure accompanied with cricoid depression; and b) assisted expiration by the release of above nose and cricoid maneuver but with simultaneous abdomen-compression. The above assisted ventilation cycle was maintained at a rate of 0-20 cycles per minute. The scopist executed both the FB and the nose-closure and release, whereas an assistant delivered the abdomen compression.
Procedure: NIV rate: 10-20/min — A basic PhO2 flow was routinely provided. A small pharyngeal catheter with warmed, humidified and fixed pure oxygen flow was inserted via one nostril to ensured catheter tip positioning in the oropharynx. The NIV was performed in the following steps. Firmly closed the mouth, then intermittently applied a) assisted inspiration by nose-closure accompanied with cricoid depression; and b) assisted expiration by the release of above nose and cricoid maneuver but with simultaneous abdomen-compression. The above assisted ventilation cycle was maintained at a rate of 0-20 cycles per minute. The scopist executed both the FB and the nose-closure and release, whereas an assistant delivered the abdomen compression.
Procedure: NIV rate: 5-10/min — A basic PhO2 flow was routinely provided. A small pharyngeal catheter with warmed, humidified and fixed pure oxygen flow was inserted via one nostril to ensured catheter tip positioning in the oropharynx. The NIV was performed in the following steps. Firmly closed the mouth, then intermittently applied a) assisted inspiration by nose-closure accompanied with cricoid depression; and b) assisted expiration by the release of above nose and cricoid maneuver but with simultaneous abdomen-compression. The above assisted ventilation cycle was maintained at a rate of 0-20 cycles per minute. The scopist executed both the FB and the nose-closure and release, whereas an assistant delivered the abdomen compression.

SUMMARY:
Introduction: The non-invasive ventilation (NIV) of continuous nasopharyngeal O2 with intermittent close/open nose and abdomen compression (PO2-NC-AC) can provide effective oxygenation, ventilation and circulation. It needs no any instruments, therefore no limits upper and lower airways. Both animal, clinical studies and experiences have already demonstrated its safety and efficacy in high risky and severe asphyxiated conditions. Making pressure (PEEP and PIP) changes is an essential for creating assist PPV. In children, airway lumen images are dynamic and positively correlate to the intraluminal pressure levels, such as the lumen open or close pressure. Closely measuring and monitoring these airway pressures and associated lumen image changes can benefit for making accurate diagnosis and enhance clinical management.

Purpose: Prospective study to evaluate the dynamic changes of upper and lower airway: 1) PEEP and PIP levels; and 2) the associated changes of lumen image by using FB with this NIV technique in small children with airway anomaly.

Study candidates: Children who: a) need FB examination or management for clinical reasons; b) age ≤5 year-old; and c) with airway anomaly; will enroll to this study. Expect enrolls a total of 30 children in one-year period.

Methods: As usually doing the FB with cardiopulmonary monitor and this NIV support in pediatric intensive care unit settings. A small catheter connects the inner cannel of FB and links to a pressure monitor. During course of FB, records the intra-airway lumen pressures (PEEP, PIP) and takes associated images. Total record (study) time in each enrolled case about 5 minutes. This study will not prolong the FB time. Finally, analysis these associated data.

Prediction: This study (30 enrolled cases) can smoothly complete in one-year period.

Benefits: This modality of FB with NIV may: 1) more safely doing; 2) get scientific data to prove it's efficacy; and 3) benefit for both clinical diagnosis and management; in children with airway anomaly.

DETAILED DESCRIPTION:
* As usually doing the FB with cardiopulmonary monitor and this NIV support in pediatric intensive care unit settings.
* A small catheter connects the inner cannel of FB and links to a pressure monitor.
* During course of FB, records the intra-lumen pressures (PEEP, PIP) and takes associated images at assigned 6 airway locations, if possible.
* These 6 locations are: Oropharynx, Supra-glottis, Mid-trachea, Supra-carina Right main bronchus, and Left main bronchus.
* Thus, a complete FB would involve 6 pairs of measurements in each child.
* Both results of PIP levels and images were then stored in a computer for later analysis.
* Total record (study) time in each enrolled case about 5 minutes. This study will not prolong the FB time. Finally, analysis these associated data.
* For objective evaluation of the lumen changes, three captured images were grouped by 6 locations in each child. These lumen dimensions were independently judged on a five-point Likert scale (1 to 5: very collapse, collapse, average, expansion, very expansion) within one week by four qualified pediatric bronchoscopists who were blinded to the source of these images. The final scores were averaged and analyzed.
* Statistical Analysis: The categorical variables were described as percentages and compared with the Chi-square or Fisher's exact test as appropriate. A two-tailed p <0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age no more than 3 years old
* a natural airway lumen without prior plasty;
* difficult weaning from current respiratory support and therefore
* scheduled for elective FB for highly suspected airway problems.

Exclusion Criteria:

* uncontrollable cardiopulmonary failure
* body weight less than 2.0 kg
* bleeding tendency.
* fixed/ too narrowed airways where the FB (OD 3.8 mm) could not pass through

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Intra- airway Positive inspiration pressure (PIP) | intra-procedure, when the tips of FB locate in the assigned airway location
  When doing these 3 modes of NIV, measure the intra-airway PIP at 6 assigned different locations.
  When doing this NIV, measure the PIP at 6 different airway locations

SECONDARY OUTCOMES:
Intra-airway lumen expansion | intra-procedure, when the tips of FB locate in the assigned airway location
  When doing these 3 modes of NIV, take and measure the lumen expansion at 6 different airway locations.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jue Soong, Study Director — University of Alberta
Locations (2):
- Taiwan (2):
  - Taipei-Veterans General Hospital, Taipei
  - Teipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided
When these data are reasonable for this study.

REFERENCES:
- [Result] Lin YT, Lee YS, Jeng MJ, Chen WY, Tsao PC, Chan IC, Soong WJ. Flexible bronchoscopic findings and the relationship to repeated extubation failure in critical children. J Chin Med Assoc. 2018 Sep;81(9):804-810. doi: 10.1016/j.jcma.2018.03.008. Epub 2018 May 31. PMID 29861210
- [Result] Soong WJ, Tsao PC, Lee YS, Yang CF. Flexible endoscopy for pediatric tracheobronchial metallic stent placement, maintenance and long-term outcomes. PLoS One. 2018 Feb 8;13(2):e0192557. doi: 10.1371/journal.pone.0192557. eCollection 2018. PMID 29420596
- [Result] Soong WJ, Tsao PC, Lee YS, Yang CF. Therapeutic flexible airway endoscopy of small children in a tertiary referral center-11 years' experience. PLoS One. 2017 Aug 17;12(8):e0183078. doi: 10.1371/journal.pone.0183078. eCollection 2017. PMID 28817604
- [Result] Soong WJ, Tsao PC, Lee YS, Yang CF. Retrieval of tracheobronchial foreign bodies by short flexible endoscopy in children. Int J Pediatr Otorhinolaryngol. 2017 Apr;95:109-113. doi: 10.1016/j.ijporl.2017.01.033. Epub 2017 Feb 16. PMID 28576517
- [Result] Soong WJ, Tsao PC, Lee YS, Yang CF, Liao J, Jeng MJ. Retrieving difficult aspirated pen caps by balloon catheter with short working-length flexible endoscopy and noninvasive ventilation support in intensive care unit. Int J Pediatr Otorhinolaryngol. 2015 Sep;79(9):1484-9. doi: 10.1016/j.ijporl.2015.06.033. Epub 2015 Jul 3. PMID 26188901
- [Result] Yang CF, Niu DM, Jeng MJ, Lee YS, Taso PC, Soong WJ. Late-onset Pompe disease with left-sided bronchomalacia. Respir Care. 2015 Feb;60(2):e26-9. doi: 10.4187/respcare.03419. Epub 2014 Oct 14. PMID 25316892
- [Result] Soong WJ, Jeng MJ, Lee YS, Tsao PC, Harloff M, Matthew Soong YH. A novel technique of non-invasive ventilation: Pharyngeal oxygen with nose-closure and abdominal-compression--Aid for pediatric flexible bronchoscopy. Pediatr Pulmonol. 2015 Jun;50(6):568-75. doi: 10.1002/ppul.23028. Epub 2014 Mar 10. PMID 24616304
- [Result] Soong WJ, Jeng MJ, Lee YS, Tsao PC, Soong YH. Nasopharyngeal oxygen with intermittent nose-close and abdomen-compression: a novel resuscitation technique in a piglet model. Pediatr Pulmonol. 2013 Mar;48(3):288-94. doi: 10.1002/ppul.22592. Epub 2012 May 2. PMID 22553182
- [Result] Soong WJ, Lee YS, Tsao PC, Yang CF, Jeng MJ. Comparison of oxygenation among different supplemental oxygen methods during flexible bronchoscopy in infants. J Chin Med Assoc. 2011 Dec;74(12):556-60. doi: 10.1016/j.jcma.2011.09.016. Epub 2011 Oct 28. PMID 22196471
- [Result] Soong WJ, Jeng MJ, Lee YS, Tsao PC, Yang CF, Soong YH. Pediatric obstructive fibrinous tracheal pseudomembrane--characteristics and management with flexible bronchoscopy. Int J Pediatr Otorhinolaryngol. 2011 Aug;75(8):1005-9. doi: 10.1016/j.ijporl.2011.04.020. Epub 2011 Jun 2. PMID 21640393
- [Result] Peng YY, Soong WJ, Lee YS, Tsao PC, Yang CF, Jeng MJ. Flexible bronchoscopy as a valuable diagnostic and therapeutic tool in pediatric intensive care patients: a report on 5 years of experience. Pediatr Pulmonol. 2011 Oct;46(10):1031-7. doi: 10.1002/ppul.21464. Epub 2011 May 27. PMID 21626712
- [Result] Soong WJ, Shiao AS, Jeng MJ, Lee YS, Tsao PC, Yang CF, Soong YH. Comparison between rigid and flexible laser supraglottoplasty in the treatment of severe laryngomalacia in infants. Int J Pediatr Otorhinolaryngol. 2011 Jun;75(6):824-9. doi: 10.1016/j.ijporl.2011.03.016. Epub 2011 Apr 21. PMID 21513991
- [Result] Soong WJ, Lee YS, Soong YH, Tsao PC, Yang CF, Jeng MJ, Peng YY. Tracheal foreign body after laser supraglottoplasty: a hidden but risky complication of an aluminum foil tape-wrapped endotracheal tube. Int J Pediatr Otorhinolaryngol. 2010 Dec;74(12):1432-4. doi: 10.1016/j.ijporl.2010.08.019. Epub 2010 Oct 8. PMID 20934755
- [Result] Chen WT, Soong WJ, Lee YS, Jeng MJ, Chang HL, Hwang B. The safety of aerodigestive tract flexible endoscopy as an outpatient procedure in young children. J Chin Med Assoc. 2008 Mar;71(3):128-34. doi: 10.1016/S1726-4901(08)70004-2. PMID 18364264
- [Result] Soong WJ. Endoscopic intubation with aid of mechanical ventilation via a dedicated nasopharyngeal airway. J Chin Med Assoc. 2007 Sep;70(9):400-2. doi: 10.1016/S1726-4901(08)70028-5. PMID 17908656
- [Result] Soong WJ. Endoscopic diagnosis and management of iatrogenic cervical esophageal perforation in extremely premature infants. J Chin Med Assoc. 2007 Apr;70(4):171-5. doi: 10.1016/S1726-4901(09)70352-1. PMID 17475599
- [Result] Soong WJ, Yuh YS. Ingested button battery retrieved by a modified magnet endoscope. J Chin Med Assoc. 2007 Mar;70(3):132-5. doi: 10.1016/S1726-4901(09)70344-2. PMID 17389159
- [Result] Yang CF, Soong WJ, Jeng MJ, Chen SJ, Lee YS, Tsao PC, Hwang B, Wei CF, Chin TW, Liu C. Esophageal atresia with tracheoesophageal fistula: ten years of experience in an institute. J Chin Med Assoc. 2006 Jul;69(7):317-21. doi: 10.1016/S1726-4901(09)70265-5. PMID 16903645
- [Result] Soong WJ. Adjusting the endotracheal tube tip in management of tracheomalacia in an infant. Int J Pediatr Otorhinolaryngol. 2004 Aug;68(8):1105-8. doi: 10.1016/j.ijporl.2004.04.001. PMID 15236902
- [Result] Lee YS, Soong WJ, Jeng MJ, Cheng CY, Shen CM, Sun J, Chen CF, Hwang B. Flexible endoscopy of aerodigestive tract in small infants. Pediatr Int. 2003 Oct;45(5):530-3. doi: 10.1046/j.1442-200x.2003.01785.x. PMID 14521526
- [Result] Lee YS, Soong WJ, Jeng MJ, Cheng CY, Shen CM, Sun J, Hwang B. Endotracheal tube position in pediatrics and neonates: comparison between flexible fiberoptic bronchoscopy and chest radiograph. Zhonghua Yi Xue Za Zhi (Taipei). 2002 Jul;65(7):341-4. PMID 12365653
- [Result] Shen CM, Soong WJ, Jeng MJ, Lee YS, Cheng CY, Sun J, Hwang B. Nasopharyngeal tract length measurement in infants. Acta Paediatr Taiwan. 2002 Mar-Apr;43(2):82-5. PMID 12041622
- [Result] Soong WJ, Jeng MJ, Hwang B. Respiratory support of children with a retropharyngeal abscess with nasal CPAP. Clin Pediatr (Phila). 2001 Jan;40(1):55-6. doi: 10.1177/000992280104000109. No abstract available. PMID 11210089
- [Result] Soong WJ, Hwang B. Intratracheal oxygen administration during bronchoscopy in newborns: comparison between two different weight groups of infants. Zhonghua Yi Xue Za Zhi (Taipei). 2000 Sep;63(9):696-703. PMID 11037646
- [Result] Soong WJ, Jeng MJ, Hwang B. The application of a modified mini-flexible-fiberoptic endoscopy in pediatric practice. Zhonghua Yi Xue Za Zhi (Taipei). 1995 Nov;56(5):338-44. PMID 8605649
- [Result] Soong WJ, Jeng MJ, Hwang B. Direct tracheobronchial suction for massive post-extubation atelectasis in premature infants. Zhonghua Min Guo Xiao Er Ke Yi Xue Hui Za Zhi. 1996 Jul-Aug;37(4):266-71. PMID 8854348
- [Result] Soong WJ, Hwang B, Tang RB. Continuous positive airway pressure by nasal prongs in bronchiolitis. Pediatr Pulmonol. 1993 Sep;16(3):163-6. doi: 10.1002/ppul.1950160305. PMID 8309740
- [Result] Soong WJ, Hwang BT. Selective placement of bronchial suction catheters in intubated full term and premature neonates. Zhonghua Yi Xue Za Zhi (Taipei). 1991 Jul;48(1):45-8. PMID 1653092
- [Result] Soong WJ, Hwang B, Deng JF, Tiu CM. New therapy for hydrocarbon pneumonitis--nasal prongs continuous positive airway pressure (NPCPAP). Zhonghua Yi Xue Za Zhi (Taipei). 1991 Jan;47(1):59-64. PMID 1848465